CLINICAL TRIAL: NCT01997814
Title: EFFECT OF SRP WITH ADJUNCTIVE THERAPY OF HERBAL IMMUNOMODULATORS ON THE SERUM C REACTIVE PROTEIN (CRP) LEVELS & CLINICAL PARAMETERS IN CHRONIC PERIODONTITIS PATIENTS - A RANDOMISED, DOUBLE BLIND, PLACEBO CONTROLLED, CLINICAL TRIAL.
Brief Title: Role of Herbal Immunomodulators in the Treatment of Chronic Periodontitis
Acronym: Septilin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tatyasaheb Kore Dental College (Other)
Responsible Party: Principal Investigator, GIRISH DEORE, Principal Investigator, Tatyasaheb Kore Dental College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TKDC12
Record Dates: First submitted 2013-11-19; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Periodontitis
Keywords: Herbal medicine,; Host modulation therapy,; Periodontitis,; Meta-analysis,; Scaling and root planing.
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — septilin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Test Group (Active Comparator): Patients in Test Group were given Herbal Immunomodulators (SeptilinTM) 2 tablets twice daily for 3 weeks then medications were stopped and changes in all parameters were again checked after 6 weeks.
  Interventions: Drug: herbal immunomodulator
- Control Group (Placebo Comparator): Patients in Control Group were given placebo drug 2 tablets twice daily for 3 weeks then medications were stopped and changes in all parameters were again checked after 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: herbal immunomodulator — Patients in Test Group were treated with scaling and root planing (SRP) along with Herbal Immunomodulators (Septilin) therapy, 2 tablets twice daily for 3 weeks.
  Other Names: Septilin (brand name)
  Arms: Test Group
Drug: Placebo — Patients in Control Group were treated with scaling and root planing (SRP) along with Placebo therapy, 2 tablets twice daily for 3 weeks.
  Arms: Control Group

SUMMARY:
Addition of systemic herbal immunomodulators with scaling & root planing (SRP) may enhance the therapeutic result of Chronic Periodontitis owing to host modulation & anti-inflammatory properties. If proven, herbal immunomodulators can be used as an adjunct to SRP.

ELIGIBILITY:
Inclusion Criteria:

1. Patients within age group of 30 to 55 years.
2. Systemically healthy individuals.
3. Patients with chronic generalized periodontitis (moderate and severe) according to Center of Disease Control (CDC) working group, 2007 criteria

Exclusion Criteria:

1. Patients with systemic illnesses (i.e., diabetes mellitus, cancer, human immunodeficiency syndrome, bone metabolic diseases, or disorders that compromise wound healing, radiation, or immunosuppressive therapy),
2. Smoking,
3. Chronic alcoholics,
4. Pregnancy or lactation,
5. Use of Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), steroids or antibiotics / antimicrobials within January 2012 to Jun 2013,
6. Confirmed or suspected intolerance to herbal medicines,
7. Periodontal therapy done within the january 2012 to Jun 2013.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in serum CRP levels at 3 weeks and 6 weeks | baseline, 3 weeks, 6 weeks
  changes from baseline in biochemical parameter, serum CRP levels were assessed at 3 weeks after starting therapy with herbal immunomodulators, then therapy was stopped and same changes were again assessed at 6 weeks from baseline. Serum CRP level was measured in milligram/liter (mg/l)
changes from baseline in Pocket Depth (PD) at 3 weeks and 6 weeks. | baseline, 3 weeks and 6 weeks
  changes from baseline in standard clinical parameter, PD were assessed at 3 weeks after starting therapy with herbal immunomodulators, then therapy was stopped and same changes were again assessed at 6 weeks from baseline. PD was measured in millimeters.
changes from baseline in Clinical Attachment Level (CAL) at 3 weeks and 6 weeks. | baseline, 3 weeks and 6 weeks
  changes from baseline in standard clinical parameter, CAL were assessed at 3 weeks after starting therapy with herbal immunomodulators, then therapy was stopped and same changes were again assessed at 6 weeks from baseline. PD was measured in millimeters.

SECONDARY OUTCOMES:
Changes from baseline in Gingival Index (GI) at 3 weeks and 6 weeks | baseline, 3 weeks and 6 weeks
  changes from baseline in standard clinical parameter, GI were assessed at 3 weeks after starting therapy with herbal immunomodulators, then therapy was stopped and same changes were again assessed at 6 weeks from baseline. GI has a scoring criteria specified by Silness & Loe, 1963.
change from baseline in Plaque Index (PI) at 3 weeks and 6 weeks | baseline, 3 weeks and 6 weeks
  changes from baseline in standard clinical parameter, PI were assessed at 3 weeks after starting therapy with herbal immunomodulators, then therapy was stopped and same changes were again assessed at 6 weeks from baseline. PI has a scoring criteria specified by Loe & Silness, 1964.
Changes from baseline in Oral Hygiene Index Simplified (OHIS) at 3 weeks and 6 weeks. | baseline, 3 weeks and 6 weeks
  changes from baseline in standard clinical parameter, OHIS were assessed at 3 weeks after starting therapy with herbal immunomodulators, then therapy was stopped and same changes were again assessed at 6 weeks from baseline. OHIS has a scoring criteria specified by Greene and Vermilion, 1964.
Changes from baseline in Sulcus Bleeding Index (SBI) at 3 weeks and 6 weeks | baseline, 3 weeks and 6 weeks
  changes from baseline in standard clinical parameter, SBI were assessed at 3 weeks after starting therapy with herbal immunomodulators, then therapy was stopped and same changes were again assessed at 6 weeks from baseline. SBI has a scoring criteria specified by Muhleman's (1971).

CONTACTS AND LOCATIONS:
Overall Officials: Girish D Deore, BDS, Principal Investigator — Post Graduate Student
Locations (1):
- Tatyasaheb Kore Dental College and Research Centre, New Pargaon, Kolhāpur, Maharashtra, India